CLINICAL TRIAL: NCT06011512
Title: Risk of Diabetes Mellitus in Patients With Giant Cell Arthritis and Polymyalgia Rheumatica.
Status: Recruiting | Type: Observational
Sponsor: Salome Kristensen (Other)
Responsible Party: Sponsor-Investigator, Salome Kristensen, MD, PhD, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: AalborgGCA
Record Dates: First submitted 2023-08-10; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Giant Cell Arteritis; Polymyalgia Rheumatica; Large Vessel Vasculitis
MeSH Terms: conditions — Giant Cell Arteritis; Polymyalgia Rheumatica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to expand the knowledge about development and aggreviation of diabetes mellitus in patients with giant cell arthritis and polymyalgia rheumatica.

The main questions it aims to answer are:

* To identify the risk of comorbidities, especially diabetes, in patients with giant cell arthritis and polymyalgia rheumatica, treated with glucocorticoids in combination with or without interleukin-6 inhibitor.
* To identify clinical outcomes and biomarkers as potential predictors for development or aggregation of already existing diabetes mellitus in patients with giant cell arthritis or polymyalgia rheumatica using machine learning prediction.

Participants will be followed at their respective rheumatology clinic, and will be asked to deliver blood samples at predefined visits.

DETAILED DESCRIPTION:
The cohort study is a prospective national cohort study in patients with giant cell arthritis (GCA) and polymyalgia rheumatica (PMR). At baseline and follow-up visits at month 1, 3, 6, 12, and every year while patients are treated at departments of rheumatology, collection of demographics, clinical data, patient reported outcomes and blood samples (Regionernes blod- og GenomBank) will occur.

Trial procedure:

Diagnostic information and referral history:

At enrollment, patients will be registered as either incident (first visit within 3 months from diagnosis) or prevalent. The patients diagnosis, time of diagnosis, type of physician establishing diagnosis, time of symptom onset, time of referral, time of first visit, date of prednisolone start, initial prednisolone dose, basis for diagnosis (clinical, classification criteria, biochemical, ultrasound, PET/CT, other imaging modalities, temporal artery biopsy), fulfillment of 1990 ACR classification criteria for GCA, fulfillment of 2018 DCVAS classification criteria for GCA, fulfillment of 2012 EULAR PMR classification criteria will be recorded. Disease stratification will be performed according to clinical diagnosis and imaging test results available. Accordingly, patients will be categorized as either 'GCA', 'PMR', 'GCA and PMR'. If a GCA diagnosis is established, patients will be further categorized as 'c-GCA', 'LV-GCA'

Clinical evaluation:

At each visit, physician disease activity category; remission, potential relapse without treatment escalation, relapse (treatment escalation, refractory disease) will be recorded. Any relapse, that lead to treatment intensification since last study visit, will be recorded. If a relapse is suspected at the current visit, the findings supporting the suspicion of disease activity and the therapeutic consequence, will be recorded.

Demography:

The patients age, gender, height, weight and history of smoking and alcohol consumption will be recorded at enrollment.

Medication:

At each visit current dose of prednisolone, methotrexate or IL-6i treatment are recorded. Date of start and discontinuation and reason for discontinuation of immunosuppressive therapy will be recorded.

Adverse events and treatment related disease burden:

Adverse effects that cause change in treatment strategy will be recorded.

DM:

At each visit data regarding development of diabetes, aggreviation of exciting DM, HgbA1c and blood glucose will be recorded.

Patient reported outcome measures (PROMs): At each visit patients will be asked to report

* Patient global numerical rang scale (NRS, 0-10)
* Patient pain NRS, neck, shoulder, pelvic, thigh (0-10)
* Patient pain NRS headache (0-10)
* Duration of morning stiffness (minutes)
* Morning stiffness NRS (0-10)
* European Quality of life -5dimension5-levels (EQ-5D-5L)

Laboratory test:

Routine blood analysis, including CRP and HbA1c, will be performed as standard of care and according to the National Danish GCA and PMR management guideline [5]. At each visit, CRP will be recorded. HbA1c and time of analysis of HbA1c can be recorded at any visit. Additionally, biobank blood samples will be collected at each study visit (study-related procedure):

* 1 × EDTA plasma tube (lavender-top), 9 ml
* 1 × Full blood DNA, 1.5 ml
* 2 × EDTA plasma, 2 ml
* 1 × EDTA buffy coat,
* 2 × serum tube (red-top), 9 ml
* 4 × serum tube, 2 ml

Time of blood sampling will be recorded. A time frame of ± 2 weeks from time of study visit will be accepted for CRP and biobank samples. However, collection of planned blood samples at any study visit, where a relapse is suspected, is strived for before treatment escalation. Furthermore, CD36, sCD36, homeostatic model assessment for insulin resistance (HOMA-IR), proinsulin C-peptide, fasting proinsulin C-peptide and fasting blood glucose are of special interest. For a subgroup of patients, oral glucose tolerance test will be performed. Biomarkers will be analysed at Aalborg University Hospital in collaboration with department of Clinical Biochemistry. Data will be gathered from Aalborg university hospital and in order to strengthen the study, further data from other departments of rheumatology will be requested from the DANIVAS database (Danish national database of patients with GCA and PMR).

Patient data can be collected at any time during their disease course.

Type of visits performed:

* Enrolment visit: First visit
* Follow up visits:
* Treatment response visit: Visits scheduled 1-2 months after treatment start or intensification to assess the effect of treatment.
* Planned follow up
* Suspected relapse or adverse events visit: An extra visit on the suspicion of relapse or adverse events potentially requiring treatment adjustment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 50 to 85 years
* Are diagnosed with GCA or PMR
* Diagnosis is established by or confirmed by a rheumatologist (clinical expert opinion)
* Speak and understand Danish
* Are able to give signed and dated informed consent

Exclusion Criteria:

* None

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population from which the cohort will be selected from, are patients who are treated at their respective outpatient rheumatology clinic. At least 8 departments of rheumatlogy in Denmark are expected to include patients.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants developing diabetes mellitus during the study period, measured in changes of HbA1c. | At baseline, and month 1, 3, 6, 12, 24 and 36.
  HbA1c is glycated hemoglobin, which means that hemoglobin is chemically bound to glucose in the bloodstream. HbA1c is a relative measure of the average glucose in the bloodstream during the past 3 months, and is used to diagnose patients with diabetes mellitus.

SECONDARY OUTCOMES:
Changes in CD36. | At baseline, and month 1, 3, 6, 12, 24 and 36.
  CD36 is a protein that helps importing fatty acids inside the cell.
Changes in sCD36. | At baseline, and month 1, 3, 6, 12, 24 and 36.
  CD36 is a protein that helps importing fatty acids inside the cell.
Changes in homeostatic model assessment for insulin resistance. | At baseline, and month 1, 3, 6, 12, 24 and 36.
  Homeostatic model assessment for insulin resistance (HOMA-IR) is a score that approximates insulin resistance.
Changes in proinsulin C-peptide. | At baseline, and month 1, 3, 6, 12, 24 and 36.
  Proinsulin C-peptide is a marker for the insulinproduction.
Changes in fasting proinsulin C-peptide. | At baseline, and month 1, 3, 6, 12, 24 and 36.
  Proinsulin C-peptide is a marker for the insulinproduction.
Changes in fasting blood glucose. | At baseline, and month 1, 3, 6, 12, 24 and 36.
  Blood glucose is the amount of glucose in the bloodstream.
Changes in CRP. | At baseline, and month 1, 3, 6, 12, 24 and 36.
  CRP is a pro-inflammatory marker.
Changes in patient pain numerical rating scale, neck, shoulder, pelvic, thigh (0-10). | At baseline, and month 12, 24, 36, 48, and 60.
  Patient pain numerical rating scale, neck, shoulder, pelvic, thigh is a rating scale in which patients are asked to rate the pain from 0 to 10 in the chosen areas, with 0 being "no pain" and 10 being "worst pain imaginable".
Changes in patient pain numerical rating scale headache (0-10). | At baseline, and month 12, 24, 36, 48, and 60.
  Patient pain numerical rating scale headache is a rating scale in which patients are asked to rate their headache pain from 0 to 10 with 0 being "no pain" and 10 being "worst pain imaginable".
Changes in duration of morning stiffness. | At baseline, and month 12, 24, 36, 48, and 60.
  With regard to duration of morning stiffness, patients are asked to rate the duration of their morning stiffness with 0 being no stiffness and 10 being 2 hours of stiffness or more.
Changes in morning stiffness numerical rating scale (0-10). | At baseline, and month 12, 24, 36, 48, and 60.
  Moring stiffness numerical rating scale is a measure of the difficulty the morning stiffness are causing, with 0 being "no difficulty" and 10 being "the worst imaginable difficulty".
Changes in European Quality of life-5dimension5-levels | At baseline, and month 12, 24, 36, 48, and 60.
  European Quality of life-5dimension5-levels is descriptive system that measures patients health related quality of life. This system consists of 5 dimensions: Mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension consists of 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
Duration and cumulative glucocorticoid dosage | At baseline, and month 1, 3, 6, 12, 24 and 36.
  It is known that treatment with glucocorticoid dosage in patients with inflammatory diseases is the number one reason for drug-induced hyperglycaemia and DM, and that GC can aggreviate hyperglycaemia in patients with a prior diagnosis of DM.

CONTACTS AND LOCATIONS:
Overall Officials: Salome Kristensen, MD, PhD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, North Denmark, Denmark